CLINICAL TRIAL: NCT02052479
Title: Differences in Insulin Secretion and Insulin Sensitivity/Resistance in African-American and Caucasian Adolescent Females With Polycystic Ovary Syndrome
Brief Title: Insulin Differences Between African-American and Caucasian Female Adolescents With Polycystic Ovary Syndrome (PCOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Rachel-Marie Cazeau, Pediatric Endocrinology Fellow, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 297013
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Polycystic Ovary Syndrome; PCOS
Keywords: Polycystic Ovary Syndrome; PCOS; Secondary Amenorrhea; Hirsutism; Hyperandrogenism; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hirsutism; Hyperandrogenism; Insulin Resistance

ARMS (2):
- Polycystic Ovary Synrome, PCOS, Caucasian, No treatment (Other): Frequently Sampled Intravenous Glucose Tolerance Test with minimal model analysis (MINMOD FSIVGTT)
  Interventions: Other: Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT)
- Polycystic Ovary Synrome, PCOS, African-American, No treatment (Other): Frequently Sampled Intravenous Glucose Tolerance Test with minimal model analysis (MINMOD FSIVGTT)
  Interventions: Other: Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT)

INTERVENTIONS:
Other: Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT)

SUMMARY:
The purpose of this research study is to see if there are differences between African-American and Caucasian girls with Polycystic Ovary Syndrome (PCOS) in how their bodies respond to a type of sugar, called glucose, the body's main source of energy. PCOS is one of the most common endocrine disorders among females. Features can include anovulation (eggs are not released from the ovaries) resulting in irregular menstrual periods, excessive amounts of androgenic (male) hormones resulting in acne and hirsutism (excessive hair growth on the face and body), and polycystic ovaries (small sac-like structures [cysts] on your ovaries) seen on ultrasound. Girls with PCOS also have higher levels of insulin in their bodies (called hyperinsulinism) but are not able to use insulin very well (called insulin resistance) resulting in an increased risk of diabetes. Diabetes is when you have high levels of glucose (sugar) in your blood. Many studies have looked at how bodies respond to glucose and have shown that compared to Caucasians, healthy African-Americans produce much more insulin (hyperinsulinism) but are not able to use it as well (insulin resistance) in childhood, adolescence, and adulthood. Insulin is a hormone that helps glucose move from the blood into the muscles for the body to use as energy. PCOS is associated with increased levels of insulin (hyperinsulinism) and not being able to use it as well (insulin resistance). So we want to see if there is a difference in insulin production (secretion) and insulin resistance between African-Americans and Caucasians girls with PCOS. To do this, we will look at blood glucose and insulin levels in response to giving glucose in African-American and Caucasian girls who have PCOS. The results of this study may ultimately help to more effectively target treatment therapy in individuals with PCOS that have increased insulin secretion and/or increased insulin resistance.

DETAILED DESCRIPTION:
PCOS is the most common endocrine abnormality of reproductive-aged women in the United States, affecting approximately 5 million women (1). The exact prevalence of PCOS in the adolescent population is unknown mainly attributed to the diagnostic challenge PCOS presents as the characteristics of normal puberty overlap with the signs and symptoms of PCOS (2). The key features of PCOS include menstrual irregularity, hyper¬androgenism, and polycystic ovarian morphology on ultrasound. However, clinical presentation may vary. It is a complex heterogeneous condition with life-long psychological, reproductive, and metabolic manifestations that impact a woman's health throughout her lifespan. PCOS is associated with major metabolic consequences including hyperinsulinism (i.e. increased insulin secretion), insulin resistance (i.e. decreased insulin sensitivity), obesity, type 2 diabetes mellitus, dyslipidemia, cardiovascular disease, endothelial dysfunction, defective fibrino¬lysis, as well as endometrial carcinoma (3).

Particular disease processes show a predilection for certain racial and ethnic groups. African-American [AA] adults are at increased risk of obesity, type 2 diabetes mellitus, cardiovascular disease mortality, and hyper¬tension compared to Caucasian [CA] adults. Past studies (4-9) have found that AAs have increased insulin secretion and decreased insulin sensitivity compared to their CA counterparts in adolescence and adulthood and even in childhood. These findings are secondary to the combination of increased insulin secretion and resistance with decreased insulin sensitivity and clearance noted in African-Americans. It is this combination of altered glucose metabolism that places AAs at increased risk of cardiovascular and metabolic morbidity. It has been proposed that hyperinsulinism or increased insulin secretion is a compensatory response by the pancreatic β-cell to increased insulin resistance. However, it has also been speculated that it is insulin resistance that is the compensatory response occurring in response to insulin hyper-secretion caused by pancreatic β-cell dysregulation (10-11).

Hyperinsulinism and insulin resistance are known inherent features of PCOS. Several studies have demonstrated significant hyperinsulinism with insulin resistance and lowered insulin sensitivity in adolescents and adults with PCOS when compared to BMI-matched healthy control subjects (12-18). Marked differences in insulin sensitivity/resistance and PCOS phenotype have been reported in adults of different races/ethnicities with PCOS (19-23), however; other studies have refuted these claims (24-27). The objective of this study is to examine the differences in insulin secretion between AA and CA adolescents with PCOS. We will also examine differences in insulin sensitivity/resistance between AA and CA adolescents with PCOS.

Primary Aim: To determine the influence of racial/ethnic background on insulin secretion in adolescent females with PCOS.

Secondary Aim: To determine the influence of racial/ethnic background on insulin sensitivity/resistance in adolescent females with PCOS.

Hypothesis: AA adolescent females with PCOS will have increased insulin secretion and decreased insulin sensitivity (i.e. increased insulin resistance) compared to CA adolescent females with PCOS.

To address this hypothesis, we will utilize one of the gold standards endorsed by the American Diabetes Association that satisfactorily assess insulin secretion and insulin sensitivity/resistance. The method utilized in this study is the frequently sampled intravenous glucose tolerance test with minimal model analysis (MINMOD FSIVGTT) (28-32). Using the data that is gathered as part of our primary and secondary aims, we will also conduct an exploratory analysis to examine the influence of PCOS phenotype on insulin secretion and insulin sensitivity/resistance and the influence of racial/ethnic background on PCOS phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents ages 12-18 years
* African-American and Caucasian females
* Menarchal for at least 2 years
* Hemoglobin A1C <6.5%
* Medical Condition: Polycystic Ovary Syndrome (PCOS) - based on AES criteria: HA in addition to ANOV and/or PCO

  * Hyperandrogenism (required): Serum Testosterone > 50 ng/dl or Free Testosterone (%) > 1.4% or Free Testosterone > 7 pg/mL
  * Oligo- and/or Anovulation: menstrual cycles lengths > 35 days and/or < 8 menstrual cycles a year
  * Polycystic Ovaries: transabdominal or trans-vaginal ultrasound finding of 12 or more follicles measuring 2-6 mm in diameter or increased ovarian volume (> 10 mL)
* Medications: Medication-naive to treatment therapy with Metformin, Oral Contraceptives, and Anti-androgen medications

Exclusion Criteria:

* Ages <12 or >18
* Prepubertal, Premenarche
* Hemoglobin A1C ≥6.5%
* Medical Conditions: Hypothyroidism, Hyperthyroidism, Diabetes Mellitus, Congenital Adrenal Hyperplasia, Hyperprolactinemia, Pregnancy
* Medications: Past and/or Present treatment therapy with Metformin, Oral Contraceptives, Anti-androgen medications, Insulin or oral hypoglycemic agents

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Insulin Secretion | -10, 0, 2, 4, 6, 8, 12, 14, 16, 19, 22, 27, 32, 42, 52, 62, 72, 82, and 92 minutes
  The objective of this study is to examine the differences in insulin secretion between AA and CA adolescents with PCOS. Primary Aim: To determine the influence of racial/ethnic background on insulin secretion in adolescent females with PCOS.

SECONDARY OUTCOMES:
Insulin Sensitivity/Resistance | -10, 0, 2, 4, 6, 8, 12, 14, 16, 19, 22, 27, 32, 42, 52, 62, 72, 82, and 92 minutes
  The objective of this study is to examine differences in insulin sensitivity/resistance between AA and CA adolescents with PCOS. Secondary Aim: To determine the influence of racial/ethnic background on insulin sensitivity/resistance in adolescent females with PCOS.

OTHER OUTCOMES:
Exploratory Analysis | -10, 0, 2, 4, 6, 8, 12, 14, 16, 19, 22, 27, 32, 42, 52, 62, 72, 82, and 92 minutes
  Using the data that is gathered as part of our primary and secondary aims, we will also conduct an exploratory analysis to examine the influence of PCOS phenotype on insulin secretion and insulin sensitivity/resistance and the influence of racial/ethnic background on PCOS phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center at The Ohio University Wexner Medical Center / Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- See also: Information on Polycystic Ovary Syndrome — http://www.hormone.org/diseases-and-conditions/womens-health/polycystic-ovary-syndrome